CLINICAL TRIAL: NCT00384865
Title: A Clinical Trial of Aspirin and Simvastatin in Pulmonary Arterial Hypertension
Brief Title: A Study of Aspirin and Simvastatin in Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 458; R01HL082895-01 (NIH)
Record Dates: First submitted 2006-09-30; First posted 2006-10-06 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Simvastatin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aspirin 81 mg + Simvastatin 40 mg (Active Comparator): Simvastatin: Simvastatin 40 mg, taken orally, once a day for 6 months
  Aspirin: Aspirin 81 mg, taken orally, once a day for 6 months
  Interventions: Drug: Simvastatin; Drug: Aspirin
- Aspirin 81 mg + Placebo (Active Comparator): Aspirin: Aspirin 81 mg, taken orally, once a day for 6 months
  Placebo taken orally, once a day for 6 months
  Interventions: Drug: Aspirin; Drug: Placebo
- Placebo + Simvastatin 40 mg (Active Comparator): Placebo taken orally, once a day for 6 months
  Simvastatin: Simvastatin 40 mg, taken orally, once a day for 6 months
  Interventions: Drug: Simvastatin; Drug: Placebo
- Placebo + Placebo (Placebo Comparator): Placebo taken orally, once a day for 6 months
  Placebo taken orally, once a day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg, taken orally, once a day for 6 months
  Other Names: Zocor
  Arms: Aspirin 81 mg + Simvastatin 40 mg; Placebo + Simvastatin 40 mg
Drug: Aspirin — Aspirin 81 mg, taken orally, once a day for 6 months
  Other Names: acetylsalicylic acid
  Arms: Aspirin 81 mg + Placebo; Aspirin 81 mg + Simvastatin 40 mg
Drug: Placebo — Placebo, taken orally, once a day for 6 months
  Arms: Aspirin 81 mg + Placebo; Placebo + Placebo; Placebo + Simvastatin 40 mg

SUMMARY:
The purpose of this study is to determine whether aspirin and simvastatin are safe and effective for the treatment of pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
PAH is characterized by dyspnea, fatigue, and lower extremity edema as a result of heart failure. In PAH, in situ thrombosis may occur in the lungs, and pulmonary endothelial dysfunction is well-recognized. As aspirin inhibits platelet aggregation, there may be value in using aspirin to treat PAH. Simvastatin has beneficial effects on blood vessels in other types of cardiovascular disease. Therefore, simvastatin may similarly benefit patients with PAH.

Participants in this study will be randomly assigned to receive 6 months of daily placebo tablets, daily aspirin and daily placebo, daily simvastatin and daily placebo, or daily aspirin and daily simvastatin in a double-blind fashion. The study will compare the safety and efficacy of aspirin to placebo and simvastatin to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Mean pulmonary artery pressure greater than 25 mm Hg at rest with a pulmonary capillary wedge pressure less than 16 mm Hg
* Diagnosis of PAH that is a) idiopathic, b) familial, or c) associated with collagen vascular disease, HIV infection, congenital systemic-to-pulmonary shunt, or former anorexigen use
* Most recent pulmonary function tests showing FEV1/FVC ratio greater than 50% AND one of the following conditions: a) total lung capacity greater than 70% predicted, or b) total lung capacity between 60% and 70% of predicted value with no more than mild patchy interstitial lung disease on high resolution computerized tomography of the chest
* Ability to perform six-minute walk testing without limitations in musculoskeletal function or coordination
* Negative pregnancy test at screening visit for women of childbearing potential
* If female, willing to use adequate form of birth control

Exclusion Criteria:

* PAH related to other etiologies
* Diagnosis of sickle cell disease
* Clinically significant untreated sleep apnea, as diagnosed by polysomnography
* Left-sided valvular disease (more than moderate mitral valve stenosis or insufficiency or aortic stenosis or insufficiency), pulmonary artery or valve stenosis, or ejection fraction less than 45% on echocardiography
* Hospitalized or acutely ill
* Kidney failure
* Initiation of PAH therapy (prostacyclin analogues, endothelin [ET]-1 receptor antagonists, phosphodiesterase [PDE]-5 inhibitors) within 3 months of study entry
* Allergy or hypersensitivity to aspirin or simvastatin
* Absolute indication for aspirin or other anti-platelet therapy
* Current treatment with statin therapy
* Inability or unwillingness to avoid non-steroidal, anti-inflammatory medications for 6 months following study entry
* Current or recent use or planned treatment with one of the following: amiodarone, cyclosporine, itraconazole, ketoconazole, erythromycin, clarithromycin, HIV protease inhibitors, nefazodone, cimetidine, danazol, large quantities of grapefruit juice (more than 1 quart daily), verapamil, fibrates, or niacin
* Peptic or duodenal ulcer diagnosed within 1 year of study entry
* Gastrointestinal bleeding within 6 months prior of study entry
* Bleeding diathesis
* History of intracranial bleeding
* Anemia (hematocrit less than 30%) at screening
* International normalized ratio (INR) greater than 3.0 at screening
* Severe thrombocytopenia (less than 75,000/L) at screening
* Hepatic transaminases greater than twice the upper limit of normal at screening
* Chronic liver disease (e.g., cirrhosis, chronic hepatitis) with portal hypertension
* Current or recent (within 6 months of study entry) chronic heavy alcohol consumption
* History of myositis
* Creatine phosphokinase (CPK) greater than 1.5 times the upper limit of normal at screening
* Abnormalities of the arm or hand or past radical mastectomy that might prevent brachial artery ultrasound
* Pregnant or breastfeeding
* Current use of another investigational drug for PAH
* Received a lung transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Kawut, MD, MS, Principal Investigator — University of Pennsylvania; David J Lederer, MD, MS, Principal Investigator — Columbia University; Reda E Girgis, MB, BCh, Principal Investigator — Johns Hopkins University; Kari E Roberts, MD, Principal Investigator — Tufts University
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts University School of Medicine, Boston, Massachusetts
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Kawut SM, Bagiella E, Lederer DJ, Shimbo D, Horn EM, Roberts KE, Hill NS, Barr RG, Rosenzweig EB, Post W, Tracy RP, Palevsky HI, Hassoun PM, Girgis RE; ASA-STAT Study Group. Randomized clinical trial of aspirin and simvastatin for pulmonary arterial hypertension: ASA-STAT. Circulation. 2011 Jun 28;123(25):2985-93. doi: 10.1161/CIRCULATIONAHA.110.015693. Epub 2011 May 18. PMID 21593252
- [Derived] Al-Naamani N, Palevsky HI, Lederer DJ, Horn EM, Mathai SC, Roberts KE, Tracy RP, Hassoun PM, Girgis RE, Shimbo D, Post WS, Kawut SM; ASA-STAT Study Group. Prognostic Significance of Biomarkers in Pulmonary Arterial Hypertension. Ann Am Thorac Soc. 2016 Jan;13(1):25-30. doi: 10.1513/AnnalsATS.201508-543OC. PMID 26501464
- [Derived] Matura LA, Ventetuolo CE, Palevsky HI, Lederer DJ, Horn EM, Mathai SC, Pinder D, Archer-Chicko C, Bagiella E, Roberts KE, Tracy RP, Hassoun PM, Girgis RE, Kawut SM. Interleukin-6 and tumor necrosis factor-alpha are associated with quality of life-related symptoms in pulmonary arterial hypertension. Ann Am Thorac Soc. 2015 Mar;12(3):370-5. doi: 10.1513/AnnalsATS.201410-463OC. PMID 25615959
- [Derived] Kawut SM, Bagiella E, Shimbo D, Lederer DJ, Al-Naamani N, Roberts KE, Barr RG, Post W, Horn EM, Tracy R, Hassoun P, Girgis R; ASA-STAT Study Group. Rationale and design of a phase II clinical trial of aspirin and simvastatin for the treatment of pulmonary arterial hypertension: ASA-STAT. Contemp Clin Trials. 2011 Mar;32(2):280-7. doi: 10.1016/j.cct.2010.12.005. Epub 2010 Dec 10. PMID 21146637

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin 81 mg + Simvastatin 40 mg | Aspirin 81 mg + Placebo | Placebo + Simvastatin 40 mg | Placebo + Placebo
Started | 16 | 16 | 16 | 16
Completed Six Month Assessment | 11 | 12 | 15 | 11
Completed | 16 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin 81 mg + Simvastatin 40 mg | Aspirin 81 mg + Placebo | Placebo + Simvastatin 40 mg | Placebo + Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (16.6) | 56.75 (13.2) | 58.6 (11.7) | 63.5 (14.2) | 59.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 15 | 14 | 55
  Male | 5 | 1 | 1 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 5 | 0 | 8
  Not Hispanic or Latino | 14 | 15 | 11 | 16 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 5 | 13
  White | 13 | 11 | 12 | 9 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 16 | 16 | 64

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked in Six Minutes
Time Frame: Measured at 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Groups:
- Aspirin 81 mg: Aspirin 81 mg, taken orally, once a day for 6 months
- Aspirin Placebo; Simvastatin Placebo: Placebo, taken orally, once a day for 6 months
- Simvastatin 40 mg: Simvastatin 40 mg, taken orally, once a day for 6 months
Arm/Group | Aspirin 81 mg | Aspirin Placebo | Simvastatin 40 mg | Simvastatin Placebo
Number analyzed (Participants) | 32 | 33 | 32 | 33
meters | 438.0 [415.9 to 460.1] | 438.5 [419.2 to 457.8] | 425.0 [400.2 to 449.9] | 452.7 [431.9 to 473.4]

2. Secondary Outcome: Time to Clinical Worsening Events (Number of Events)
Description: Defined by the addition of new PAH therapies or dose increases in previously stable PAH therapy, hospitalization for right-sided heart failure, lung transplantation, atrial septostomy, and cardiovascular and all-cause death.
Time Frame: Measured at 6 months
Measure: Number; unit: events
Arm/Group | Aspirin 81 mg | Aspirin Placebo | Simvastatin 40 mg | Simvastatin Placebo
Number analyzed (Participants) | 32 | 33 | 32 | 33
events | 2 | 6 | 4 | 4

3. Secondary Outcome: Adverse Events
Description: Please refer to the Adverse Event Tables for specific information
Time Frame: Measured at 6 months
Measure: Number; unit: events
Arm/Group | Aspirin 81 mg | Aspirin Placebo | Simvastatin 40 mg | Simvastatin Placebo
Number analyzed (Participants) | 32 | 33 | 32 | 33
events | 59 | 66 | 66 | 58

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each subject from screening through 6 months after enrollment/randomization
Arm/Group | Aspirin 81 mg | Aspirin Placebo | Simvastatin 40 mg | Simvastatin Placebo
Serious Adverse Events (participants affected / at risk) | 4/32 | 1/33 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 32/32 | 33/33 | 32/32 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin 81 mg (N=32) | Aspirin Placebo (N=33) | Simvastatin 40 mg (N=32) | Simvastatin Placebo (N=33)
Major Bleeding Episode (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin 81 mg (N=32) | Aspirin Placebo (N=33) | Simvastatin 40 mg (N=32) | Simvastatin Placebo (N=33)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11) | 12 (12) | 9 (9)
Bruising (General disorders) | 8 (8) | 8 (8) | 10 (10) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 3 (3) | 5 (5)
Headache (General disorders) | 5 (5) | 3 (3) | 5 (5) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3) | 4 (4)
Other Infections (Infections and infestations) | 4 (4) | 4 (4) | 4 (4) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (2)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
Increased Transaminases (Hepatobiliary disorders) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Insomnia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Minor Bleeding Episode (Blood and lymphatic system disorders) | 11 (11) | 12 (12) | 14 (14) | 13 (13)

LIMITATIONS AND CAVEATS:
* The primary end point that should be used in early-stage clinical trials in PAH is uncertain.
* We did not include invasive hemodynamic end points.
* Early termination led to missing data for those active subjects in the trial at termination (n16).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No